CLINICAL TRIAL: NCT05718596
Title: The Antimicrobial Efficacy of Sweeps Laser Compared to Ultrasonically Activated Irrigation and Needle Irrigation in Posterior Teeth With Apical Periodontitis: A Clinical Study
Brief Title: Quantitative Assessment of the Efficacy of Sweeps Laser Activation Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seyda Ersahan, DDS, PhD (Other)
Responsible Party: Sponsor-Investigator, Seyda Ersahan, DDS, PhD, The Antimicrobial Efficacy of Sweeps Laser Compared to Ultrasonically Activated Irrigation and Needle Irrigation in Posterior Teeth With Apical Periodontitis: A Clinical Study, Istanbul Medipol University Hospital
Organization: Istanbul Medipol University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Microbial analysis root canal
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Periapical Periodontitis; Polymerase Chain Reaction; Enterococcus Faecalis Infection
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sweeps laser (Experimental): use of sweeps laser irrigation activation
  Interventions: Other: sweeps laser to use irrigation activation
- pasif ultrasonic irrigation (PUI) (Experimental): Pasif ultrasonic irrigation (PUI) -VDW Ultra
  Interventions: Other: PUI to use irrigation activation

INTERVENTIONS:
Other: sweeps laser to use irrigation activation — The SWEEPS fiber tip (25 µs ultra-short dual pulse mode-Auto SWEEPS mode) was inserted into the Er:YAG laser source (2,940 nm, 20 mJ per pulse, 15 Hz, 0.3 W power, and 50 µs pulse frequency). 3% NaOCl solution was activated in three periods of 20 s. Then, the same procedure was repeated with 2 ml of 17% EDTA solution.
  Arms: Sweeps laser
Other: PUI to use irrigation activation — The irrigation solution was used by adapting an ultrasonic tip (IRRI S 21/25; VDW, Munich, Germany) to an ultrasonic device (VDW Ultra; VDW, Munich, Germany). The tip was activated a total of three times, with each cycle lasting 20 s and involving the use of 1 ml of 3% NaOCl. Then, 2 ml of 17% EDTA solution was activated for 1 min as describe above. The ultrasonic tip was placed 2 mm behind the working length without touching the canal walls.
  Arms: pasif ultrasonic irrigation (PUI)

SUMMARY:
Aim of the present study was to determine the intraradicular microbiota of previously root canal-treated teeth with apical periodontitis using droplet digital polymerase chain reaction (ddPCR) and to investigate the antibacterial effectiveness of different irrigation activation methods [ Sweeps laser and PUI group ] that will make classical chemomechanical preparation more effective. This superiority, parallel, randomized clinical trial was conducted in the clinic of the Endodontic Department, Faculty of Dentistry, Istanbul Medipol University, Istanbul. 30 patients with apical periodontitis (one tooth each) were randomly allocated into two groups according to the used (n=15, for each): the Sweeps laser group (A) or the vdw ultra group (B). Total bacterial loads, as well as the amount of Enterococcus faecalis (E.faecalis) were determined before (S1) and after (S2) chemomechanical preparation and finally, after intracanal medication (S3) by means of ddPCR.

DETAILED DESCRIPTION:
Eligibility criteria The study population consisted of 30 patients (aged 19-66 years) presenting to the endodontic clinic at Istanbul Medipol University Dental School, for nonsurgical endodontic treatment of teeth with apical periodontitis lesions. 30 teeth exhibiting clinical and radiographic evidence of chronic apical periodontitis lesions were included in this study. BT lab branded ELISA Kits (Shangai, China) were used to measure IL-1Beta levels. Radiographically, the diameter of the periapical radiolucency ranged from 2 to 7 mm. Teeth with apical periodontitis had required treatment. Selected teeth had enough crown structure for adequate isolation with a rubber dam and showed an absence of periodontal pockets or attachment level deeper than 4 mm. Exclusion criteria were also applied, as follows: teeth from patients who had received antibiotics within the previous 3 months or who had any general disease, teeth that could not be properly isolated with rubber dam, teeth with absence of coronary sealing, teeth with periodontal pocket depth >4 mm; and teeth with crown/root fracture. Only one tooth was included from each patient.

Root canal treatment procedures and sampling Rubber dam and an aseptic technique were used throughout the endodontic retreatment. After plaque removal and rubber dam isolation, the operative field was cleaned with 3% hydrogen peroxide and disinfected with 2.5% NaOCl solution. Then, all coronal restorations, posts and carious defects were removed and access preparation was completed when the root canal filling was properly exposed. Afterwards, the tooth (including the pulp chamber), clamp, and adjacent rubber dam were once again disinfected with 2.5% NaOCl, followed by inactivation with 10% sodium thiosulfate in order to avoid interference with bacteriological sampling. Sterility control samples (SR1) were taken from the tooth surface with a sterile Omni Swab (Whatman FTA, Sigma-Aldrich) with an ejectable head. Paper points were transferred to cryotubes containing phosphate buffered saline (PBS) solution stored at -20°C. In each case, a single root canal was sampled in order to confine the microbial evaluation to a single ecological environment. In multirooted teeth, the root with the periapical lesion was selected. If there were periapical lesions in all roots, the wider canal was selected.

The working length (WL) was established 1-mm short of the apical foramen with an apex locator (Raypex6; VDW GmbH, Munich, Germany), and then periapical radiographs were taken to ensure that all filling material was removed. Irrigation with sterile saline solution was performed in order to remove any remaining materials and to moisten the canal prior to sample collection. Next, the canal was left filled with saline, and a small hand instrument was placed at the WL and used to gently file the canal walls. An initial microbiologic sample (S1) was taken from the root canal with sterile paper points consecutively placed at the WL. Three sterile paper points were inserted into the root canal for sampling. Each paper point was left in the canal for about 1 minute. Both the paper points and the endodontic hand instrument, without the handle, were transferred to cryotubes containing 300 μl of PBS solution stored at -20°C. The samples were transferred to genetic analysis laboratory for further analysis in cold chain.

Root canals were prepared by using the ProTaper Next; Dentsply-Sirona, Ballaigues, İsviçre files and irrigated with 2.5% NaOCl. The canals were apically enlarged to size 35 (AS35) at the working length. Between each instrument change, the root canal was irrigated with 5 ml of 2.5% NaOCl solution by using 30-gauge side-vented needle, which was placed 1 to 2 mm short of working length. Hence, a total of 30 mL of the irrigating solution was used. After instrumentation was completed, the smear layer was removed with 2 mL 17% EDTA, which was left in the canal for 3 min, followed by 2.5% NaOCl. The root canal was dried with sterile paper points and flushed with 2 ml of 10% sodium thiosulfate for 1 min to inactivate the NaOCl solution. Next, a sample (S2) was taken from the canals as described for S1. Following this, the NaOCl was agitated/activated as described below.

Sweeps group: The SWEEPS fiber tip (25 µs ultra-short dual pulse mode-Auto SWEEPS mode) was inserted into the Er:YAG laser source (2,940 nm, 20 mJ per pulse, 15 Hz, 0.3 W power, and 50 µs pulse frequency). The SWEEPS tip placed in the access cavity was kept in a stable position, and activation was performed in the SWEEPS mode using the same method with the same amount of irrigation solutions described for the PIPS group.

PUI group: The irrigation solution was used by adapting an ultrasonic tip (IRRI S 21/25; VDW, Munich, Germany) to an ultrasonic device (VDW Ultra; VDW, Munich, Germany). The tip was activated a total of three times, with each cycle lasting 20 s and involving the use of 1 ml of 3% NaOCl. Then, 2 ml of 17% EDTA solution was activated for 1 min as describe above. The ultrasonic tip was placed 2 mm behind the working length without touching the canal walls.

Finally, the canals in both groups were dried and rinsed with 2 mL 10% sodium thiosulfate for 1 min. The post activation sample (S3) was obtained in the same way as the pre-activation sample was collected and sent for the PCR analysis. Completion of the root canal treatment proceeded with root filling using lateral condensation of gutta-percha. Access cavities were restored with composite resin, and a final radiograph was taken. All the root canal and microbial sampling procedures were performed by a single experienced endodontist. Total bacterial loads, as well as the amount of Enterococcus faecalis were determined before instrumentation, after instrumentation and use of the irrigation activation systems, by means of droplet digital polymerase chain reaction (ddPCR).

Total bacterial loads, as well as the amount of Enterococcus faecalis were determined before instrumentation, after instrumentation and use of the intracanal medicaments, by means of ddPCR.

Genomic DNA isolation and measurement of DNA concentration DNA was extracted using the QIAamp DNA Mini Kit (Qiagen, Germany) following the protocol recommended by the manufacturer. Before DNA isolation, samples (the tubes with paper points) were digested at 50-60°C BY vortexING for 30s in every 10 min in order to ensure disaggregation of all bacteria into the PBS solution. Afterwards, the paper points were aseptically removed from the suspension and, the bacterial suspension was pelleted by centrifugation for 10 min at 5000 g. The pellet was then resuspended in 180 µl buffer ATL supplied by QIAamp DNA Mini Kit (QIAGEN GmbH, Hilden, Germany) and 20 µl proteinase K (20 mg/ml) was added. Samples were incubated for 3 h at 56°C. Subsequently, total bacterial genomic DNA was isolated according to the protocol of the QIAamp DNA Mini Kit. The final volume of DNA solution of each sample was 150 μL and was taken into account during calculation. DNA concentration (absorbance at 260 nm) was determined with a spectrophotometer (Promega Quantifluor).

Amplification of 16S rRNA genes Primers for Universal and Enterococcus 16S rRNA genes were designed in this study. After DNA extraction of samples with QIAamp DNA Mini Kit, 700-800 bp of 16S rRNA sequences were amplified by using universal E8F forward primer (5'-AGAGTTTGATCCTGGCTCAG-3') and universal E1115R reverse primer (5'-AGGGTTGCGCTCGTTG-3') 59. The final volume of PCR reactions for each isolated bacterial strain was adjusted to 25 µl. The amplification reactions of 16S rRNA genes were performed with the following conditions. 1 cycle of predenaturation at 95°C for 3 minutes, 35 cycles of 95°C for 30 seconds, 55°C for 30 seconds, and 72°C for 30 seconds which continue with a final extension step at 72°C for 10 minutes.

The PCR products were analyzed by electrophoresis using 2% agarose gel (containing ethidium bromide) in Tris/BoratE/EDTA (TBE) buffer, with gels being analyzed under ultraviolet light (at 140V for 20 minutes). Their images were visualized under ultraviolet illumination. In addition, the control and optimization of primers to be used for ddPCR was also done in conventional PCR.

Purification and Sequencing of the 16S rRNA Gene After the PCR reactions, the purification of PCR products is done by hydrolyzing the excess primers and nucleotides with ExoSap-IT (Thermo, PN: 78201.1.ML) containing Exonuclease I and Alkaline Phosphatase enzymes. 2 µl of ExoSap-IT was mixed with 5 µl of PCR product for each sample. The ExoSap reaction is performed at 37 °C for 15 minutes (enzyme activation) followed by 15 minutes (inactivation) at 80 °C. Sequencing reactions were performed by using Bigdye™ Terminator v3.1 cycle sequencing kit (Thermo). The reactions were performed according to the kit manual for all isolated strains.

After purification of the products with Exosap, the sequence reaction was performed with BigDye Terminator v3.1 Cycle Sequencing Kit (Thermo) under the following conditions. After the sequence PCR, BigDye products were purified by colon method. Zymo ZR DNA Sequencing Clean-up Kit (Zymo Research, USA) was used for this process. All samples were purified in accordance with the protocol given in the kit and executed on the 3130XL genetic analyzer.

Droplet Digital PCR (ddPCR) Droplet Digital PCR (ddPCR) was performed using primers designed according to the 16S rRNA region specific to the total bacteria and Enterococcus faecalis species, after sequencing, absolute quantitation from the bacterial species found in the paper-point sample. Primer pairs were 16S-F-5'-AGGGAATCTTCSGCAATGGG-3' and 16S-R-5'-ACGCCCAATAAATCCGGACA-'3 for total bacteria and ENT-F-5'-CGCTTCTTTCCTCCCGAGT-3' and ENT-R-5'-GCCATGCGGCATAAACTG-3' primer pairs for Enterococcus Faecalis. In the PCR reaction, amplicons amplified with unmarked primer pairs were analyzed by labeling with Eva-Green dye. For absolute quantitation of Enterococcus and total 16S rRNA, PCR was performed with two primer pairs from the same sample. 20 µL of PCR mix containing 10 µL of 2X ddPCR EvaGreen Supermix (Bio-Rad, cat. no. 1864034), 9 µL of nuclease-free water, 0.25 µL of both forward and reverse primer and 2 ng of DNA from each sample Thermal cycling conditions were: 95◦C for 5 min, then 40 cycles of 95◦C for 30 s and 60◦C for 1 min and two final steps at 4◦C for 5 minutes and 90◦C for 5minutes with a 4◦C infinite hold. After PCR was completed, the sealed plate was transferred into the plate holder of the QX200 Droplet Reader (Bio-Rad, cat. no. 1864003).

ELIGIBILITY:
Inclusion Criteria:

* root canal-treated teeth exhibiting clinical and radiographic evidence of chronic apical periodontitis lesions.
* Teeth with lesion apical periodontitis
* Radiographically, the diameter of the periapical radiolucency ranged from 2 to 7 mm.
* The teeth had intact coronal restorations, with no obvious exposure of the root-filling material to the oral cavity.
* Selected teeth had enough crown structure for adequate isolation with a rubber dam and showed an absence of periodontal pockets or attachment level deeper than 4 mm.

Exclusion Criteria:

* teeth from patients who had received antibiotics within the previous 3 months or who had any general disease, teeth that could not be properly isolated with rubber dam, teeth with absence of coronary sealing, teeth with periodontal pocket depth >4 mm; and teeth with crown/root fracture. Only one tooth was included from each patient.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-10 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
the sequence analysis of 16S rRNA genes by the Sanger sequencing | hrough study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: SEYDA ERSAHAN, Assoc.Prof., Principal Investigator — IstanbulMedipol University
Locations (1):
- Istanbul Medipol University, Faculty of Dentistry, Istanbul, Esenler, Turkey (Türkiye)